CLINICAL TRIAL: NCT02025569
Title: The Effectiveness of Strain Counterstrain in the Treatment of Patients With Chronic Ankle Instability: a Randomized Clinical Trial
Brief Title: The Effect of Strain-counterstrain on Ankle Instability
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Data collection was terminated due to unavailability of additional participants.
Sponsor: Long Island University (Other)
Responsible Party: Principal Investigator, Cristiana Kahl Collins, PT, PhD, Assistant Professor, Long Island University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CKCollins-SCS
Record Dates: First submitted 2013-12-24; First posted 2014-01-01 (Estimated); Last update posted 2014-01-01 (Estimated); Status verified 2013-12

CONDITIONS: Other Instability, Ankle and Foot
Keywords: chronic ankle instability; lateral ankle sprain; manual therapy; star excursion balance test; strain and counterstrain
MeSH Terms: conditions — Sprains and Strains

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental group (Experimental): Strain counterstrain intervention
  Interventions: Other: Strain Counterstrain
- Control Group (Sham Comparator): Sham Strain Counterstrain intervention
  Interventions: Other: Sham strain counterstrain

INTERVENTIONS:
Other: Strain Counterstrain
  Arms: Experimental group
Other: Sham strain counterstrain
  Arms: Control Group

SUMMARY:
This study seeks to determine the effectiveness of Strain Counterstrain in the treatment of chronic ankle instability.

DETAILED DESCRIPTION:
This study aimed to determine the effect of Strain Counterstrain (SCS) on dynamic balance and subjective sense of instability in individuals with chronic ankle instability (CAI). Although many studies have been published on CAI, the cause for this common clinical dysfunction remains inconclusive. No studies have assessed the effectiveness of SCS on CAI. Baseline information on all participants includes a demographic questionnaire, the Star Excursion Balance Test (SEBT), and the Foot and Ankle Ability Measure (FAAM). Participants were randomized into the SCS intervention group or the sham SCS control group. All participants received an intervention (as assigned) once a week for four weeks in addition to performing a prescribed home exercise program. At week four all participants repeated the outcome measures and completed a Global Rating of Change (GROC) form. The primary aim was examined with a 2-way analysis of variance (ANOVA).

ELIGIBILITY:
Inclusion Criteria:

* history of at least 1 ankle sprain, with pain and/or limping for more than 1 day, at least 3 months earlier
* 3 of more episodes of ankle giving way in the last 12 months
* chronic instability attributed to the original sprain injury
* age between 18-55

Exclusion Criteria:

* history of fracture or surgery in the affected ankle
* any other lower extremity musculoskeletal injury on the side of the involved ankle
* vestibular dysfunction or disorder
* history of balance dysfunction
* history of stroke or any other neurological pathology or disease
* history of ACL injury
* current participation in physical therapy or rehabilitation for the ankle injury
* evidence of CNS dysfunction

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2008-01; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Star Excursion Balance Test | baseline
  A measure assessing dynamic standing balance as the individual stands on one leg and reaches, with the other leg, in eight different directions. The distances reached with the non-stance leg are measured.
Star Excursion Balance Test | 4 weeks
  A measure assessing dynamic standing balance as the individual stands on one leg and reaches, with the other leg, in eight different directions. The distances reached with the non-stance leg are measured.

SECONDARY OUTCOMES:
Foot and Ankle Ability Measure | baseline
  This measures assesses ankle function skills subjectively via a questionnaire
Foot and Ankle Ability Measure | 4 weeks
  This measures assesses ankle function skills subjectively via a questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Cristiana K Collins, PhD, Principal Investigator — Long Island University
Locations (1):
- Long Island University, Brooklyn, New York, United States